CLINICAL TRIAL: NCT01742364
Title: A Randomized Clinical Trial in Adults and Newborns to Compare the Safety, Reactogenicity and Immunogenicity of BCG Administration Via a Disposable Syringe Jet Injector (DSJI) to BCG Administration Via Syringe and Needle
Brief Title: Comparative Study of Bacille Calmette Guerin (BCG) Delivery Via Disposable Syringe Jet Injector and Needle & Syringe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: World Health Organization (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS 645
Record Dates: First submitted 2012-11-30; First posted 2012-12-05 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2013-12

CONDITIONS: Tuberculosis
Keywords: disposable syringe jet injector (DSJI); DSJI; BCG; tuberculosis; intradermal delivery; South Africa
MeSH Terms: conditions — Tuberculosis | interventions — Needles; Syringes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bioject Intradermal (ID) Pen (Experimental): Intradermal administration of BCG vaccine via the Bioject ID Pen.
  Interventions: Device: Bioject ID Pen
- Needle and syringe (Active Comparator): Intradermal administration of BCG vaccine via needle and syringe.
  Interventions: Device: Needle and syringe

INTERVENTIONS:
Device: Bioject ID Pen — Participants in this arm will receive a standard dose of BCG via the Bioject ID needle-free jet injector device (investigational administration technique).
  Other Names: Disposable Syringe Jet Injector; DSJI; Jet Injector; ID Pen
  Arms: Bioject Intradermal (ID) Pen
Device: Needle and syringe — Participants in this arm will receive a standard dose of BCG via syringe and needle by the Mantoux technique (standard of care administration technique).
  Arms: Needle and syringe

SUMMARY:
The study is designed to test the hypothesis that BCG administration via jet injector will produce a comparable immune response and that there will be no significant differences in safety or reactogenicity between BCG administration via jet injector and needle and syringe.

The primary objectives of this study are to...

1. Compare the safety and reactogenicity of BCG administered intradermally by a jet injector device in adults and infants, to BCG administered intradermally by needle and syringe;
2. Compare the specific T cell immunity in neonates vaccinated with BCG via the jet injector device to infants vaccinated with BCG via needle and syringe.

DETAILED DESCRIPTION:
A randomized, controlled, partially blinded clinical trial in 2 stages (adult stage, infant stage) will be applied at a single site.

The first stage will include thirty (30) adult participants. The Data Safety Monitoring Board (DSMB) will evaluate the reactogenicity and safety data for all 30 adults up to day 28 after vaccination. Pending a favourable safety review by the DSMB, the second stage in sixty-six (66) newborn participants will commence. Potential adult and infant participants will be screened prior to enrolment to apply inclusion and exclusion criteria.Note that as the adult stage was a pilot, only results of the infant study are presented here.

In each of the stages half of the study population (15 adults, 33 neonates) will receive BCG via conventional syringe and needle (standard of care administration technique), and half (15 adults, 33 neonates) will receive BCG via jet injector (investigational administration technique). A single and standard volume and dose of BCG will be administered per the package insert. Neonates will receive their BCG shortly after birth.

The occurrence of injection site reactogenicity events and systemic adverse events will be compared between study groups in both adults and neonates. In the neonate stage, BCG and M.tb specific immunogenicity will also be compared between study groups.

For the adult stage the vaccinator and participant will be unblinded to study arm allocation. For the infant stage, the vaccinator will be unblinded but the participant caregiver will be blinded. For both the adult and infant stages the follow-up team will be blinded to study arm allocation. The laboratory will be blinded to study arm allocation for the infant stage immunogenicity assays.

The trial will be conducted at the field site of the South African Tuberculosis Vaccine Initiative (SATVI) in the Cape Winelands East district of the Western Cape of South Africa. Recruitment and vaccination of neonates will take place at 1 or more of the state public healthcare antenatal clinics and birthing units in the area. Recruitment and vaccination of adults, as well as follow-up of adults and the neonates/infants will take place on the SATVI field site premises, or on the premises of the public healthcare clinic. All study procedures, including vaccination, will be performed by SATVI study staff.

ELIGIBILITY:
Adult stage

* Inclusion criteria:

  1. Male or female, age 18 to 50 years.
  2. Written informed consent, including permission for access to medical records and an HIV test.
  3. Available for study follow up and display a willingness and capacity to comply to study procedures.
  4. In good general health, as assessed by medical history and a focused physical examination.
  5. HIV test (rapid test, ELISA [enzyme-linked immunosorbent assay], or PCR [polymerase chain reaction]) negative.
  6. Quantiferon®-TB Gold (Cellestis) test for latent TB infection negative within 2 weeks of enrolment.
  7. BCG vaccination at birth as confirmed by history or the presence of a BCG scar.
  8. In the case of female participants, a negative urine or serum pregnancy test at enrolment, and not pregnant or lactating. Evidence of contraception is not required since BCG is not contra-indicated in pregnancy.
* Exclusion criteria:

  1. A history or evidence of a significant or chronic medical condition or disease.
  2. Skin condition, bruising or birth mark at the intended injection site.
  3. History of previous active tuberculosis (TB) disease or current active TB disease.
  4. History of a household contact with active TB disease who has received less than 2 months treatment.

Neonate Stage

* Inclusion criteria:

  1. Male or female neonates within 48 hours of birth.
  2. Written informed consent, including permission to access medical records and results of antenatal HIV tests.
  3. Infant participants and their caregivers available for study follow-up and display the willingness and capacity to comply with study procedures.
  4. Neonates must be in good general health as assessed by medical history during pregnancy and delivery, and focused physical examination.
  5. Birth weight more than or equal to 2500 grams.
  6. Apgar score at 5 minutes more than or equal to 7.
  7. A maternal HIV test result (rapid test, ELISA or PCR) taken during pregnancy must be available, documented and negative.
* Exclusion criteria:

  1. Participant must not have received BCG vaccination prior to enrolment.
  2. Significant antenatal or intrapartum complications that may affect the health of the neonate.
  3. Skin condition, bruising or birth mark at the intended injection site.
  4. Maternal HIV test (rapid test, ELISA or PCR) not performed antenatally, HIV test results not available, or HIV test result known positive.
  5. Maternal history of current active TB, or other household contact with known active TB disease who has received less than 2 months of treatment.

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hennie Geldenhuys, Principal Investigator — South African Tuberculosis Vaccine Initiative
Locations (1):
- SATVI, University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants: 131 consents obtained; 50 screening failures, no participation refusals, and 66 enrolled at birth. 15 infants were consented, screened, and eligible for participation but were not enrolled because the enrollment target had been reached.
  Adults: 95 consents obtained; 63 screening failures, 2 participation refusals, and 30 enrolled.
Groups:
- INFANTS: Bioject Intradermal (ID) Pen; ADULTS: Bioject Intradermal (ID) Pen: Intradermal administration of BCG vaccine via the Bioject ID Pen.
  Bioject ID Pen
- INFANTS: Needle and Syringe; ADULTS: Needle and Syringe: Intradermal administration of BCG vaccine via needle and syringe.
  Needle and syringe
Period: Overall Study
Arm/Group | INFANTS: Bioject Intradermal (ID) Pen | INFANTS: Needle and Syringe | ADULTS: Bioject Intradermal (ID) Pen | ADULTS: Needle and Syringe
Started | 33 | 33 | 15 | 15
Completed | 33 | 33 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Infants (n=66) and Adults (n=30)
Groups:
- Total: Total of all reporting groups
Arm/Group | INFANTS: Bioject Intradermal (ID) Pen | INFANTS: Needle and Syringe | ADULTS: Bioject Intradermal (ID) Pen | ADULTS: Needle and Syringe | Total
Number analyzed (Participants) | 33 | 33 | 15 | 15 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 33 | 0 | 0 | 66
  Between 18 and 65 years | 0 | 0 | 15 | 15 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 18 | 16 | 13 | 10 | 57
  Male | 15 | 17 | 2 | 5 | 39

OUTCOME MEASURES:

1. Primary Outcome: Injection Site Adverse Events (Following Injection)
Description: Injection site adverse events including redness, swelling, induration, tenderness, ulceration, fluctuation , drainage, laceration, bruising, and scarring will be monitored for up to fourteen weeks following vaccination.
Time Frame: 14 weeks
Measure: Number; unit: Adverse events
Arm/Group | INFANTS: Bioject Intradermal (ID) Pen | INFANTS: Needle and Syringe | ADULTS: Bioject Intradermal (ID) Pen | ADULTS: Needle and Syringe
Number analyzed (Participants) | 33 | 33 | 15 | 15
Adverse events | 138 | 141 | 126 | 146
Statistical Analysis 1: Comparison: INFANTS: Bioject Intradermal (ID) Pen vs INFANTS: Needle and Syringe; Comparison of all adverse events (both injection site and systemic AEs); Test type: Superiority or Other; p = 0.475, Fisher Exact
Statistical Analysis 2: Comparison: ADULTS: Bioject Intradermal (ID) Pen vs ADULTS: Needle and Syringe; Comparison of all adverse events (both injection site and systemic AEs); Test type: Superiority or Other; p = 0.187, Fisher Exact

2. Primary Outcome: Systemic Adverse Events
Description: Systemic adverse events, solicited and unsolicited, including symptoms of lethargy, disrupted feeding patterns, fever, lymphadenopathy, rash, or any other physical abnormalities will be monitored for up to fourteen weeks following vaccination.
Time Frame: 14 weeks
Measure: Number; unit: Adverse events
Groups:
- Bioject Intradermal (ID) Pen; ADULTS: Bioject Intradermal (ID) Pen: Intradermal administration of BCG vaccine via the Bioject ID Pen.
  Bioject ID Pen
Arm/Group | Bioject Intradermal (ID) Pen | INFANTS: Needle and Syringe | ADULTS: Bioject Intradermal (ID) Pen | ADULTS: Needle and Syringe
Number analyzed (Participants) | 33 | 33 | 15 | 15
Adverse events | 20 | 20 | 18 | 27

3. Primary Outcome: Short Term Whole Blood Intracellular Cytokine Staining Assay for BCG-specific CD4 (Cluster of Differentiation 4) T-cells
Description: BCG-specific immunogenicity was tested in infants only, since they are the target study population and BCG immunogenicity in adults is known to be different from that in infants.
  Utilizing a whole-blood intracellular cytokine staining (ICS) assay, we analyzed cytokine co-expression patterns by BCG-specific CD4 and CD8 T-cells. Briefly, 0.5 ml heparinized whole blood was incubated for 12 hours with BCG, no antigen or phytohemagglutinin (PHA) in the presence of anti-CD28 and anti-CD49d, with the last 5 hours including Brefeldin A prior to treating with BD FACS™ Lysing Solution and cryopreservation. Cells were batch-thawed, permeabilized with BD Perm/Wash™ buffer, and stained with fluorescent antibodies. At least 120,000 CD3+CD4+ T-cells were acquired for the no-antigen and BCG samples on a BD™ LSR II flow cytometer.
Time Frame: 10 weeks post-vaccination
Population: Due to failed phlebotomy on 5 infants, results were not available for 2 participants in the Bioject ID Pen arm and for 3 participants in the Needle and syringe arm.
  Immunogenicity was not measured for adults in the study.
Measure: Median (Inter-Quartile Range); unit: percentage responding to cytokines
Arm/Group | INFANTS: Bioject Intradermal (ID) Pen | INFANTS: Needle and Syringe
Number analyzed (Participants) | 31 | 30
percentage responding to cytokines | 0.664 [0.410 to 1.160] | 0.485 [0.308 to 0.842]
Statistical Analysis 1: Comparison: INFANTS: Bioject Intradermal (ID) Pen vs INFANTS: Needle and Syringe; Test type: Superiority or Other; p = 0.205, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Short Term Whole Blood Intracellular Cytokine Staining Assay for BCG-specific CD4 T-cells
Description: as for outcome 3
Time Frame: 14 weeks post-vaccination
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: percentage responding to cytokines
Arm/Group | INFANTS: Bioject Intradermal (ID) Pen | INFANTS: Needle and Syringe
Number analyzed (Participants) | 31 | 30
percentage responding to cytokines | 0.386 [0.242 to 0.637] | 0.325 [0.227 to 0.427]
Statistical Analysis 1: Comparison: INFANTS: Bioject Intradermal (ID) Pen vs INFANTS: Needle and Syringe; Test type: Superiority or Other; p = 0.325, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Diameter of Skin Bleb
Time Frame: Immediately post-vaccination
Measure: Number; unit: participants
Arm/Group | INFANTS: Bioject Intradermal (ID) Pen | INFANTS: Needle and Syringe | ADULTS: Bioject Intradermal (ID) Pen | ADULTS: Needle and Syringe
Number analyzed (Participants) | 33 | 33 | 15 | 15
participants
  No wheal | 0 | 12 | 0 | 0
  Wheal > 0 mm | 33 | 21 | 15 | 15
Statistical Analysis 1: Comparison: INFANTS: Bioject Intradermal (ID) Pen vs INFANTS: Needle and Syringe; Test type: Superiority or Other; p = 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: ADULTS: Bioject Intradermal (ID) Pen vs ADULTS: Needle and Syringe; Test type: Superiority or Other; p = 0.130, Kruskal-Wallis

6. Other Pre Specified Outcome: Fluid Leakage on Skin at Injection Site
Time Frame: Immediately post-vaccination
Population: For adults, the skin fluid deposition was estimated and categorized by the vaccinator (e.g., no wetness, damp skin, flow on skin, spray in air); for infants, volume was measured objectively and categorized by the filter paper technique (units in µl).
Measure: Number; unit: participants
Arm/Group | INFANTS: Bioject Intradermal (ID) Pen | INFANTS: Needle and Syringe | ADULTS: Bioject Intradermal (ID) Pen | ADULTS: Needle and Syringe
Number analyzed (Participants) | 33 | 33 | 15 | 15
participants
  ≤ 2.5 µl | 5 | 28 | 0 | 0
  > 2.5 µl to ≤ 5 µl | 12 | 2 | 0 | 0
  > 5 µl to ≤ 10 µl | 14 | 1 | 0 | 0
  > 10 µl to ≤ 20 µl | 2 | 2 | 0 | 0
  > 20 µl | 0 | 0 | 0 | 0
  No wetness | 0 | 0 | 0 | 7
  Damp skin | 0 | 0 | 15 | 8
  Flow on skin | 0 | 0 | 0 | 0
  Spray in air | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: INFANTS: Bioject Intradermal (ID) Pen vs INFANTS: Needle and Syringe; Test type: Superiority or Other; p = 0.001, Chi-squared
Statistical Analysis 2: Comparison: ADULTS: Bioject Intradermal (ID) Pen vs ADULTS: Needle and Syringe; Test type: Superiority or Other; p = 0.003, Chi-squared

ADVERSE EVENTS:
Time Frame: 14 weeks for infants, 12 weeks for adults
Description: Infants attended study visits 4, 10, and 14 weeks after vaccination, and parents were contacted by telephone 1, 7, and 14 days after vaccination. Adults were seen 1, 2, 4, and 12 weeks after vaccination.
Arm/Group | INFANTS: Bioject Intradermal (ID) Pen | INFANTS: Needle and Syringe | ADULTS: Bioject Intradermal (ID) Pen | ADULTS: Needle and Syringe
Serious Adverse Events (participants affected / at risk) | 1/33 | 4/33 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 30/33 | 27/33 | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFANTS: Bioject Intradermal (ID) Pen (N=33) | INFANTS: Needle and Syringe (N=33) | ADULTS: Bioject Intradermal (ID) Pen (N=15) | ADULTS: Needle and Syringe (N=15)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2) | 0 | 0
Viral pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
Neonatal jaundice (Endocrine disorders) | 0 | 1 (1) | 0 | 0
Urinary tract infection (Endocrine disorders) | 0 | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFANTS: Bioject Intradermal (ID) Pen (N=33) | INFANTS: Needle and Syringe (N=33) | ADULTS: Bioject Intradermal (ID) Pen (N=15) | ADULTS: Needle and Syringe (N=15)
Scar (Skin and subcutaneous tissue disorders) | 24 (24) | 17 (17) | 15 (15) | 13 (13)
Erythema (Skin and subcutaneous tissue disorders) | 30 (30) | 24 (24) | 14 (14) | 15 (17)
Ulceration (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (11) | 15 (15) | 15 (15)
Scaling (Skin and subcutaneous tissue disorders) | 6 (6) | 16 (16) | 9 (9) | 11 (11)
Pustule (Skin and subcutaneous tissue disorders) | 14 (14) | 13 (13) | 7 (7) | 7 (7)
Papule (Skin and subcutaneous tissue disorders) | 9 (9) | 9 (9) | 2 (2) | 2 (2)
Scab (Skin and subcutaneous tissue disorders) | 12 (12) | 7 (7) | 1 (1) | 3 (3)
Swelling (Skin and subcutaneous tissue disorders) | 30 (30) | 27 (27) | 1 (1) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6) | 1 (1) | 0 (0)
Diaper rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Tenderness (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 15 (16) | 15 (17)
Induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 15 (15) | 15 (17)
Drainage (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8) | 11 (11) | 14 (14)
Headache (General disorders) | 0 (0) | 0 (0) | 8 (8) | 10 (10)
Myalgia (General disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
Fatigue (General disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Pigmentation (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (5) | 0 (0) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Oral herpes zoster (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coryza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Drinking less than usual (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less